CLINICAL TRIAL: NCT01908296
Title: Phase I Study of FK949E - A Study of Drug-drug Interactions Between FK949E and Fluvoxamine in Healthy Male Adults
Brief Title: Study to Evaluate the Effect of Multiple-dose of Fluvoxamine on the Plasma Concentration of Quetiapine (FK949E) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6949-CL-0004
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy; Pharmacokinetics of Quetiapine
Keywords: FK949E; fluvoxamine; Antipsychotic; Quetiapine
MeSH Terms: interventions — Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FK949E group (Experimental): receiving FK949E with and without fluvoxamine
  Interventions: Drug: FK949E; Drug: fluvoxamine

INTERVENTIONS:
Drug: FK949E — Oral
  Other Names: extended release formulation of quetiapine
Drug: fluvoxamine — Oral
  Other Names: Luvox®

SUMMARY:
The objective of the study was to assess the effect of multiple-dose fluvoxamine on the pharmacokinetics of quetiapine (FK949E) in healthy adult male subjects. The safety of FK949E in the population was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Body weight : ≥50.0 kg, <80.0 kg
* Body Mass Index : ≥17.6, <26.4
* Healthy, as judged by the investigator/subinvestigator based on the results of physical examinations (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital admission to immediately before study medication

Exclusion Criteria:

* Subjects with the following history.

  1. Hepatic disease (e.g. viral hepatitis, drug-induced liver injury).
  2. Heart disease (e.g. congestive heart failure, angina pectoris, arrhythmia requiring

     treatment).
  3. Respiratory disease (e.g. serious bronchial asthma, chronic bronchitis)
  4. Gastrointestinal disease (e.g. serious peptic ulcer, gastroesophageal reflux esophagitis;

     diseases requiring several selections except for appendicitis)
  5. Renal disease (e.g. acute renal failure, glomerulonephritis, interstitial nephritis).
  6. Cerebrovascular disorder (e.g. cerebral infarction).
  7. Malignant tumor.
  8. Drug allergies. Allergic disorders (except for hay fever)
  9. Drug dependence, alcohol dependence
* Any disease (except dental caries)
* A deviation from the normal reference range of blood pressure, pulse rate, body temperature, or 12-lead ECG
* A deviation of the following criteria for clinical laboratory tests.

The normal reference ranges specified at the study site will be used as the normal reference ranges in the present study.

1. Hematology:

   * A deviation of ±20% from the upper or lower limit of the normal range
2. Blood biochemistry:

   * A deviation from the normal range for AST, ALT, creatinine (Cre), HbA1c or serum electrolytes.
   * A deviation of ±20% from the upper or lower limit of the normal range for other items than the above.
   * However, the lower limit of the normal range will not be established for items for which a deviation from the lower limit is not considered clinically significant[AST, ALT, total bilirubin (T-Bil), ALP, γ-GTP, LDH, CK, Cre, uric acid (UA), BUN, and total cholesterol (T-Cho)].
3. Urinalysis:

   * U-Glc and/or U-Pro results of (±) or worse
   * U-Uro results of (+) or worse
4. Urinary drug test:

   * A positive result for phencyclidine, benzodiazepine, cocaine, amphetamines, cannabis, opiates, barbiturates or tricyclic antidepressants
5. Immunological test:

   * A positive result for hepatitis B, hepatitis C, syphilis, or HIV

     * History of treatment, including medication, within 14 days before the start of study drug administration
     * Consumption of food or beverages containing St. John's Wort within 14 days before the start of study drug administration, or consumption of grapefruit
     * Previous participation in a pre- or post-marketing clinical study of another prescription drug or a medical device within 120 days before the study
     * History of administration of quetiapine
     * History of administration of fluvoxamine
     * Whole blood sampling of 400 mL or more within 90 days before the screening assessment, whole blood sampling of 200 mL or more within 30 days before the screening assessment, or blood component donation within 14 days before the screening assessment
     * Routine excessive alcohol consumption ("excessive alcohol" is defined as an average of 45 g of alcohol per day [cf., a large bottle of beer containing 25 g of alcohol, 180 mL of sake containing 22 g of alcohol])
     * Subjects with a smoking habit (except those who quit smoking at least 90 days before the screening assessment)

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of unchanged quetiapine | For 48 hours after dosing.
AUC (area under the curve) of unchanged quetiapine | For 48 hours after dosing.

SECONDARY OUTCOMES:
tmax of plasma concentration of unchanged quetiapine | For 48 hours after dosing.
t1/2 of plasma concentration of unchanged quetiapine | For 48 hours after dosing.
Maximum plasma concentration (Cmax) of quetiapine metabolites | For 48 hours after dosing.
AUC (area under the curve) of quetiapine metabolites | For 48 hours after dosing.
tmax of plasma concentration of quetiapine metabolites | For 48 hours after dosing.
t1/2 of plasma concentration of quetiapine metabolites | For 48 hours after dosing.
Maximum plasma concentration (Cmax) of unchanged fluvoxamine | For 12 hours after dosing.
AUC (area under the curve) of unchanged fluvoxamine | For 12 hours after dosing.
tmax of plasma concentration of unchanged fluvoxamine | For 12 hours after dosing.
t1/2 of plasma concentration of unchanged fluvoxamine | For 12 hours after dosing.
Safety assessed by the incidence of adverse events, clinical tab tests, vital signs, 12-lead ECGs and physical exam | Up to 20 Days.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=173